CLINICAL TRIAL: NCT04316793
Title: Neurophysiological, Biomechanical and Clinical Effects of Dry Needling Versus Sham Needling When Applied to the Infraspinatus Muscle in People With Chronic Shoulder Pain: a Randomized Pilot Study
Brief Title: Effects of Dry Needling When Applied to the Infraspinatus Muscle in People With Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Ordre Professionnel de la Physiothérapie du Québec (OPPQ) (Unknown); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nathaly Gaudreault, Full Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-3133
Record Dates: First submitted 2020-03-11; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Trigger Point Pain, Myofascial; Chronic Shoulder Pain
Keywords: Dry needling; Infraspinatus; Neurophysiological effects
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (DN) (Experimental): Intramuscular insertion
  Interventions: Other: Dry needling
- Sham needling (SN) (Sham Comparator): Intradermal insertion
  Interventions: Other: Sham needling (SN)

INTERVENTIONS:
Other: Dry needling — Intramuscular insertion of an OPTIMED 40mm x 0.3mm acupuncture needle in a trigger point of the infraspinatus muscle
  Arms: Dry needling (DN)
Other: Sham needling (SN) — Intradermal insertion of an OPTIMED 40mm x 0.3mm acupuncture needle over the infraspinatus region
  Arms: Sham needling (SN)

SUMMARY:
Up to 77% of patients with chronic shoulder pain have a trigger point (TrP) in the infraspinatus muscle. These TrPs can lead to pain, limitation of activities and reduced quality of life. Dry needling (DN) is gaining popularity as a treatment for TrPs in physiotherapy. However, its clinical effects remain poorly understood mechanistically and its neurophysiological effects little studied.

The primary objective of this study is to determine the feasibility of a larger scale study.

The secondary objective of this study is to to explore the immediate neurophysiological, biomechanical and clinical effects of DN and sham needling when applied to TrP of the infraspinatus muscle in people with chronic non-traumatic shoulder pain.

DETAILED DESCRIPTION:
Methodology

In this randomized, double-blind, parallel-group trial, twenty adults with chronic non-traumatic shoulder pain and with a infraspinatus TrP will be recruited according to established criteria. Participants will be randomized into two groups: one group (n = 10) receiving a DN in the infraspinatus TrP and another group (n = 10) receiving a sham needling.

Recruitment strategies

Recruitment will be done through posters that will be posted on bulletin boards of the Faculty of Medicine and Health Sciences of the University of Sherbrooke and in physiotherapy clinics in the region. The persons interested will be invited to contact the research assistant in charge of the study to verify their eligibility to participate.

Data collection procedure

The experimental procedure will take place in a laboratory located at the Research Center on Aging in Sherbrooke, Quebec, Canada. Upon arrival, individuals will be greeted by a research assistant. Verification of the presence of TrP in the infraspinatus to confirm eligibility to participate will be carried out by a physiotherapist with more than 20 years of experience in the identification of TrPs and with the application of DN, according to the following procedure: Participants will be asked to lie in a decubitus lateral position on a treatment table and on the asymptomatic side. The upper arm will be supported on a box placed in front of them, so that the muscles can be relaxed, but the arm will be positioned in a and have a slight horizontal adduction to slightly stretch the fibers of the infraspinatus muscle. Manual palpation with flat fingers and perpendicular to the fibers will be used to identify the tight muscle band. Once a tight muscle band has been identified, the physiotherapist will search within this band for a contraction node, namely the TrP. Once she had identified this TrP with a non-toxic black Sharpie pencil, she will validate with the patient that the compression of this TrP reproduces local or referred pain. This pain should correspond to the pain patterns known to the infraspinatus according to Simons and Travell, 1999 and reproduce the pain known by the patient. This pain should be at least a 1/10 intensity on the visual analog scale (VAS). Ineligible participants will receive advices from the physiotherapist as well as a prescription for exercises related to their condition and a list of physiotherapists they can consult.

The research assistant will explain the nature of the project to the selected participants, he will make sure that the participants have no contraindications to receive DN and/or for transcranial magnetic stimulation (TMS) examination, and he will obtain written informed consent. Participants will then complete a questionnaire used to collect baseline medical information.

Intervention (DN and Sham)

DN will be performed by a certified clinician, experienced with the technique. She will explain the purpose of the intervention and she will review the contraindications and precautions for DN to ensure that the procedure is safe. The technique used is recommended by l'Ordre professionnel de la physiothérapie du Québec (OPPQ). The clinician will insert a sterile disposable acupuncture needle, OPTIMED (non-silicone), 40 mm x 0.30 caliber. The direction of the needle will be slightly oblique, directly in the TrP and in the direction of the muscle fibers. The production of a twitch is expected, gliding and rotation of the needle may be performed to produce this effect, if necessary. The needle will be removed after the twitch. The same procedure will be used for the sham group, except that the needle will be inserted at the subcutaneous level, at the depth of the superficial adipous tissues

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral, chronic non-traumatic shoulder pain (VAS ≥ 2/10; >3 months)
2. Localized pain in the shoulder region or referred according to the territory of the infraspinatus (Travell and Simons, 1999)
3. Presence of a palpable nodule inside a tight muscle band reproducing the patient's pain

Exclusion Criteria:

1. Cancer or metastasis in organs or tissues above the pelvis (< 5 years)
2. Shoulder capsulitis
3. Shoulder, thorax or mastectomy surgeries
4. Shoulder bone fracture (< 6 months)
5. C4-C5 or C6 radiculopathy
6. Osteoporosis or excessive atrophy of the infraspinous fossa (infraspinatus <10 mm)
7. Body mass index (BMI) > 28

Exclusion (TMS security):

1. Pregnant woman
2. Neurological, psychiatric or epilepsy conditions
3. Implants (e.g. Neurostimulator, pacemaker, cerebral aneurysm clip, screw or plate), metallic foreign body in the eye
4. Head trauma with loss of consciousness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 10 months
  Average number of participants recruited per month
Exclusion rate | Through study completion, an average of 10 months
  Number of participants excluded from the study due to eligibility criteria (e.g. too narrow, are they clear)
Refusal rate | Through study completion, an average of 10 months
  Number of participants who refused to participate (e.g. fear of needle, fear of transcranial magnetic stimulation)
Retention rate | Baseline, immediately after and 24 hours post-treatment evaluation
  Number of loss at follow-up
Length of time of the procedure | Baseline, immediately after and 24 hours post-treatment evaluation
  Average time needed per participant (testing and intervention)
Safety of the procedure: adverse effects | Immediately after intervention to 24 hours post-treatment
  Listing of any adverse effects

SECONDARY OUTCOMES:
Corticospinal excitability of the infraspinatus | At baseline, immediately after intervention, 24 hours after the intervention
  Tested with transcranial magnetic stimulation (TMS) connected to a neuronavigation device, characterized by the active motor threshold and expressed in stimulator maximum power percentage
Glenohumeral arthrokinematics | At baseline, immediately after intervention, 24 hours after the intervention
  Captured images are taken using ultrasound imaging (GE Logiq-e; linear array 5-12MHz) at 0° and 30° of external rotation. Measurements in cm included: 1) subacromial space (position of the humeral head relative to the acromion); 2) anteroposterior position of the humeral head relative to the glenoid.
Pressure pain perceived | At baseline, immediately after intervention, 24 hours after the intervention
  Obtained using an algometer (directly applied on the TrP; average of three measurements taken at 30 sec. interval), characterized by the threshold of discomfort and expressed in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly Gaudreault, PhD, Study Director — Université de Sherbrooke; Mélanie Morin, PhD, Study Director — Université de Sherbrooke; Guillaume Léonard, PhD, Study Director — Université de Sherbrooke
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bron C, Franssen J, Wensing M, Oostendorp RA. Interrater reliability of palpation of myofascial trigger points in three shoulder muscles. J Man Manip Ther. 2007;15(4):203-15. doi: 10.1179/106698107790819477. PMID 19066669
- [Background] Tough EA, White AR, Richards S, Campbell J. Variability of criteria used to diagnose myofascial trigger point pain syndrome--evidence from a review of the literature. Clin J Pain. 2007 Mar-Apr;23(3):278-86. doi: 10.1097/AJP.0b013e31802fda7c. PMID 17314589
- [Background] Cagnie B, Barbe T, De Ridder E, Van Oosterwijck J, Cools A, Danneels L. The influence of dry needling of the trapezius muscle on muscle blood flow and oxygenation. J Manipulative Physiol Ther. 2012 Nov-Dec;35(9):685-91. doi: 10.1016/j.jmpt.2012.10.005. PMID 23206963
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Alonso-Blanco C, Ge HY, Arendt-Nielsen L, Arroyo-Morales M. Muscle trigger points and pressure pain hyperalgesia in the shoulder muscles in patients with unilateral shoulder impingement: a blinded, controlled study. Exp Brain Res. 2010 May;202(4):915-25. doi: 10.1007/s00221-010-2196-4. Epub 2010 Feb 26. PMID 20186400
- [Background] Rathbone ATL, Grosman-Rimon L, Kumbhare DA. Interrater Agreement of Manual Palpation for Identification of Myofascial Trigger Points: A Systematic Review and Meta-Analysis. Clin J Pain. 2017 Aug;33(8):715-729. doi: 10.1097/AJP.0000000000000459. PMID 28098584
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Arias-Buria JL, Fernandez-de-Las-Penas C, Palacios-Cena M, Koppenhaver SL, Salom-Moreno J. Exercises and Dry Needling for Subacromial Pain Syndrome: A Randomized Parallel-Group Trial. J Pain. 2017 Jan;18(1):11-18. doi: 10.1016/j.jpain.2016.08.013. Epub 2016 Oct 5. PMID 27720812
- [Background] Baldry P. The integration of acupuncture within medicine in the UK--the British Medical Acupuncture Society's 25th anniversary. Acupunct Med. 2005 Mar;23(1):2-12. doi: 10.1136/aim.23.1.2. PMID 15844434
- [Background] Cagnie B, Dewitte V, Coppieters I, Van Oosterwijck J, Cools A, Danneels L. Effect of ischemic compression on trigger points in the neck and shoulder muscles in office workers: a cohort study. J Manipulative Physiol Ther. 2013 Oct;36(8):482-9. doi: 10.1016/j.jmpt.2013.07.001. Epub 2013 Aug 28. PMID 23993756
- [Background] Chen JT, Chung KC, Hou CR, Kuan TS, Chen SM, Hong CZ. Inhibitory effect of dry needling on the spontaneous electrical activity recorded from myofascial trigger spots of rabbit skeletal muscle. Am J Phys Med Rehabil. 2001 Oct;80(10):729-35. doi: 10.1097/00002060-200110000-00004. PMID 11562554
- [Background] Dorsher PT. Can classical acupuncture points and trigger points be compared in the treatment of pain disorders? Birch's analysis revisited. J Altern Complement Med. 2008 May;14(4):353-9. doi: 10.1089/acm.2007.0810. PMID 18576919
- [Background] Fricton JR, Kroening R, Haley D, Siegert R. Myofascial pain syndrome of the head and neck: a review of clinical characteristics of 164 patients. Oral Surg Oral Med Oral Pathol. 1985 Dec;60(6):615-23. doi: 10.1016/0030-4220(85)90364-0. PMID 3865133
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Langevin HM, Churchill DL, Cipolla MJ. Mechanical signaling through connective tissue: a mechanism for the therapeutic effect of acupuncture. FASEB J. 2001 Oct;15(12):2275-82. doi: 10.1096/fj.01-0015hyp. PMID 11641255
- [Background] Langevin HM, Bouffard NA, Badger GJ, Churchill DL, Howe AK. Subcutaneous tissue fibroblast cytoskeletal remodeling induced by acupuncture: evidence for a mechanotransduction-based mechanism. J Cell Physiol. 2006 Jun;207(3):767-74. doi: 10.1002/jcp.20623. PMID 16511830
- [Background] Lucas KR, Rich PA, Polus BI. Muscle activation patterns in the scapular positioning muscles during loaded scapular plane elevation: the effects of Latent Myofascial Trigger Points. Clin Biomech (Bristol). 2010 Oct;25(8):765-70. doi: 10.1016/j.clinbiomech.2010.05.006. Epub 2010 Jul 27. PMID 20667633
- [Background] Lund I, Lundeberg T. Are minimal, superficial or sham acupuncture procedures acceptable as inert placebo controls? Acupunct Med. 2006 Mar;24(1):13-5. doi: 10.1136/aim.24.1.13. PMID 16618044
- [Background] Shah JP, Gilliams EA. Uncovering the biochemical milieu of myofascial trigger points using in vivo microdialysis: an application of muscle pain concepts to myofascial pain syndrome. J Bodyw Mov Ther. 2008 Oct;12(4):371-384. doi: 10.1016/j.jbmt.2008.06.006. Epub 2008 Aug 13. PMID 19083696
- [Background] Shah JP, Phillips TM, Danoff JV, Gerber LH. An in vivo microanalytical technique for measuring the local biochemical milieu of human skeletal muscle. J Appl Physiol (1985). 2005 Nov;99(5):1977-84. doi: 10.1152/japplphysiol.00419.2005. Epub 2005 Jul 21. PMID 16037403
- [Background] Bradnam L, Shanahan EM, Hendy K, Reed A, Skipworth T, Visser A, Lennon S. Afferent inhibition and cortical silent periods in shoulder primary motor cortex and effect of a suprascapular nerve block in people experiencing chronic shoulder pain. Clin Neurophysiol. 2016 Jan;127(1):769-778. doi: 10.1016/j.clinph.2015.03.012. Epub 2015 Apr 4. PMID 25900020
- [Background] Bradnam LV, Stinear CM, Lewis GN, Byblow WD. Task-dependent modulation of inputs to proximal upper limb following transcranial direct current stimulation of primary motor cortex. J Neurophysiol. 2010 May;103(5):2382-9. doi: 10.1152/jn.01046.2009. Epub 2010 Mar 10. PMID 20220073
- [Background] Ngomo S, Mercier C, Roy JS. Cortical mapping of the infraspinatus muscle in healthy individuals. BMC Neurosci. 2013 Apr 24;14:52. doi: 10.1186/1471-2202-14-52. PMID 23617624
- [Background] Roberts LV, Stinear CM, Lewis GN, Byblow WD. Task-dependent modulation of propriospinal inputs to human shoulder. J Neurophysiol. 2008 Oct;100(4):2109-14. doi: 10.1152/jn.90786.2008. Epub 2008 Aug 20. PMID 18715892
- [Background] Alisauskiene M, Truffert A, Vaiciene N, Magistris MR. Transcranial magnetic stimulation in clinical practice. Medicina (Kaunas). 2005;41(10):813-24. PMID 16272828
- [Background] Barker AT, Jalinous R, Freeston IL. Non-invasive magnetic stimulation of human motor cortex. Lancet. 1985 May 11;1(8437):1106-7. doi: 10.1016/s0140-6736(85)92413-4. No abstract available. PMID 2860322
- [Background] Berth A, Pap G, Neuman W, Awiszus F. Central neuromuscular dysfunction of the deltoid muscle in patients with chronic rotator cuff tears. J Orthop Traumatol. 2009 Sep;10(3):135-41. doi: 10.1007/s10195-009-0061-7. Epub 2009 Aug 19. PMID 19690944
- [Background] Brown SH, Brookham RL, Dickerson CR. High-pass filtering surface EMG in an attempt to better represent the signals detected at the intramuscular level. Muscle Nerve. 2010 Feb;41(2):234-9. doi: 10.1002/mus.21470. PMID 19722252
- [Background] Cowey A. The Ferrier Lecture 2004 what can transcranial magnetic stimulation tell us about how the brain works? Philos Trans R Soc Lond B Biol Sci. 2005 Jun 29;360(1458):1185-205. doi: 10.1098/rstb.2005.1658. PMID 16147516
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Moseley GL, Flor H. Targeting cortical representations in the treatment of chronic pain: a review. Neurorehabil Neural Repair. 2012 Jul-Aug;26(6):646-52. doi: 10.1177/1545968311433209. Epub 2012 Feb 13. PMID 22331213
- [Background] Ngomo S, Leonard G, Moffet H, Mercier C. Comparison of transcranial magnetic stimulation measures obtained at rest and under active conditions and their reliability. J Neurosci Methods. 2012 Mar 30;205(1):65-71. doi: 10.1016/j.jneumeth.2011.12.012. Epub 2011 Dec 29. PMID 22227444
- [Background] Ngomo S, Mercier C, Bouyer LJ, Savoie A, Roy JS. Alterations in central motor representation increase over time in individuals with rotator cuff tendinopathy. Clin Neurophysiol. 2015 Feb;126(2):365-71. doi: 10.1016/j.clinph.2014.05.035. Epub 2014 Jun 21. PMID 25043198
- [Background] Romero JR, Ramirez DM, Aglio LS, Gugino LD. Brain mapping using transcranial magnetic stimulation. Neurosurg Clin N Am. 2011 Apr;22(2):141-52, vii. doi: 10.1016/j.nec.2010.11.002. PMID 21435567
- [Background] Rossini PM, Rossi S. Transcranial magnetic stimulation: diagnostic, therapeutic, and research potential. Neurology. 2007 Feb 13;68(7):484-8. doi: 10.1212/01.wnl.0000250268.13789.b2. PMID 17296913
- [Derived] Laramee A, Leonard G, Morin M, Roch M, Gaudreault N. Neurophysiological and psychophysical effects of dry versus sham needling of the infraspinatus muscle in patients with chronic shoulder pain: a randomized feasibility study. Arch Physiother. 2021 Oct 18;11(1):23. doi: 10.1186/s40945-021-00118-x. PMID 34663474